CLINICAL TRIAL: NCT03868631
Title: Muscle Growth and Development Following a 12-week Resistance Training Program in Men and Women Consuming Soy and Whey Protein Supplements
Brief Title: Muscle Growth Following a Resistance Training Program in Men and Women Consuming Protein Supplements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Point Loma Nazarene University (Other)
Responsible Party: Principal Investigator, Heidi Lynch, Assistant Professor, Point Loma Nazarene University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 01435225
Record Dates: First submitted 2019-02-25; First posted 2019-03-11 (Actual); Results first posted 2020-02-27 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Skeletal Muscle Growth

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Soy protein group (Active Comparator)
  Interventions: Dietary Supplement: Soy protein supplement
- Whey protein group (Active Comparator)
  Interventions: Dietary Supplement: Whey protein supplement

INTERVENTIONS:
Dietary Supplement: Whey protein supplement — 19 g whey protein isolate (contains 2 g leucine) was consumed daily by one intervention group.
  Arms: Whey protein group
Dietary Supplement: Soy protein supplement — 26 g soy protein isolate (contains 2 g leucine) was consumed daily by the other intervention group.
  Arms: Soy protein group

SUMMARY:
Soy and whey protein have different concentrations of leucine, an amino acid known to be a particularly potent simulator of muscle protein synthesis. The purpose of this study is to determine whether matching soy and whey protein supplements for leucine content instead of by total protein content would contribute to differences in strength increases and muscle growth in response to 12 wk of resistance training.

ELIGIBILITY:
Inclusion Criteria:

* non-smoking
* body mass index (BMI) 18.5-24.9
* recreationally active

Exclusion Criteria:

* participated in structured weight training during the previous 12 month
* vegetarian or vegan
* presence of chronic disease
* pregnant, postpartum up to six months, lactating, or intention to become pregnant
* allergy to whey or soy
* changes in body weight more than 10 pounds in the past three months

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2016-08-15 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Lynch, PhD, Principal Investigator — Point Loma Nazarene University
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 282 people responded to the screening survey online from August 2016 through January 2017. Data collection was completed by May 2017. 61 participants were randomized for study participation. Recruitment emails were sent to students at Arizona State University and others were contacted via word of mouth.
Period: Baseline to Week 6
Arm/Group | Soy Protein Group | Whey Protein Group
Started | 30 | 31
Completed | 26 | 27
Not Completed | 4 | 4
Not completed — Adverse Event | 0 | 3
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 3 | 0
Period: Week 6 to Week 12 (Study Completion)
Arm/Group | Soy Protein Group | Whey Protein Group
Started | 26 | 27
Completed | 22 | 26
Not Completed | 4 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Soy Protein Group | Whey Protein Group | Total
Number analyzed (Participants) | 30 | 31 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.83 (4.27) | 22.22 (3.38) | 22.03 (3.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 21 | 42
  Male | 9 | 10 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: White | 21 | 18 | 39
  Ethnicity: Non-white | 9 | 13 | 22
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 31 | 61
Height [Mean (Standard Deviation); unit: centimeters] | 166.93 (10.03) | 168.20 (7.04) | 167.57 (8.59)
Weight [Mean (Standard Deviation); unit: kilograms] | 65.5 (13.3) | 66.9 (10.1) | 66.26 (11.61)
Lean body mass [Mean (Standard Deviation); unit: kilograms] | 44.084 (10.2896) | 44.486 (8.7167) | 44.301 (9.3816)
Appendicular lean body mass [Mean (Standard Deviation); unit: kilograms] | 19.81796 (5.353628) | 20.32806 (5.096195) | 20.09263 (5.171179)
Fat mass [Mean (Standard Deviation); unit: kilograms] | 19.71463 (6.818858) | 20.21259 (6.261987) | 19.97825 (6.468543)
Body fat percent [Mean (Standard Deviation); unit: percent body fat] | 30.92083 (8.227645) | 31.38214 (8.163188) | 31.16923 (8.115504)
Vastus lateralis thickness [Mean (Standard Deviation); unit: centimeters] | 2.167615 (0.3136369) | 2.330765 (0.5032904) | 2.253989 (0.4286374)
Vastus intermedius thickness [Mean (Standard Deviation); unit: centimeters] | 1.563921 (0.3433793) | 1.572045 (0.4095149) | 1.568222 (0.3761121)
Peak torque doing leg extensions (60 d/s) [Mean (Standard Deviation); unit: Newton-meters] | 132.0228 (44.87827) | 124.3479 (39.91502) | 127.8901 (42.03202)
Peak torque doing leg flexions (60 d/s) [Mean (Standard Deviation); unit: Newton-meters] | 64.2884 (15.04077) | 60.4792 (15.85495) | 62.2373 (15.45260)

OUTCOME MEASURES:

1. Primary Outcome: Lean Body Mass Change
Description: assessed using dual energy x-ray absorptiometry (DEXA) scan for changes in lean body mass (kg)
Time Frame: Post-12 week intervention
Measure: Mean (Standard Deviation); unit: kilogram
Arm/Group | Soy Protein Group | Whey Protein Group
Number analyzed (Participants) | 30 | 31
kilogram | 1.5 (0.4) | 1.3 (0.3)
Statistical Analysis 1: Comparison: Soy Protein Group vs Whey Protein Group; Between-group differences at baseline were compared using independent t-tests. Multilevel models for change (MLM) were used to determine differences between groups over time for study outcomes. Age, sex, and number of sessions missed were included as covariates. Time and time by group interactions were examined. Analyses were conducted using IBM SPSS Statistics version 23. Significance was set at p<0.05; Test type: Superiority; p < 0.05, multilevel models for change

2. Primary Outcome: Muscle Tissue Thickness Change
Description: assessed using changes in muscle thickness assessed by ultrasound (cm)
Time Frame: Post-12 week intervention
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | Soy Protein Group | Whey Protein Group
Number analyzed (Participants) | 30 | 31
centimeter | 0.12 (0.16) | 0.05 (0.41)

3. Primary Outcome: Leg Girth Changes
Description: assessed using circumference measurements (cm)
Time Frame: Post-12 week intervention
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | Soy Protein Group | Whey Protein Group
Number analyzed (Participants) | 30 | 31
centimeter | -0.1865 (0.05254) | -0.0084 (0.06227)

4. Secondary Outcome: Change in Peak Torque When Doing Leg Extensions
Description: Assessed using an isokinetic dynamometer set at 60 degrees of motion per second (d/s)
Time Frame: Post-12 week intervention
Measure: Mean (Standard Deviation); unit: Newton-meters
Arm/Group | Soy Protein Group | Whey Protein Group
Number analyzed (Participants) | 30 | 31
Newton-meters | 12.1 (13.5) | 18.0 (16.1)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Soy Protein Group | Whey Protein Group
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/31
Other Adverse Events (participants affected / at risk) | 2/30 | 3/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Soy Protein Group (N=30) | Whey Protein Group (N=31)
Hip pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Week 6-week 12
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — Baseline-week 6
Vomited (Gastrointestinal disorders) | 0 (0) | 1 (1) — Baseline-week 6
Knee pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Baseline-week 6
Knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Week 6-week 12

LIMITATIONS AND CAVEATS:
1. No non-protein control (ex: placebo, maltodextrin)
2. No objective measurement of physical activity outside of the exercise intervention
3. No objective verification if the participants consumed protein powder on non-training days

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2016-08-01): https://cdn.clinicaltrials.gov/large-docs/31/NCT03868631/Prot_004.pdf
  • Statistical Analysis Plan (2016-08-01): https://cdn.clinicaltrials.gov/large-docs/31/NCT03868631/SAP_005.pdf
  • Informed Consent Form (2017-01-27): https://cdn.clinicaltrials.gov/large-docs/31/NCT03868631/ICF_006.pdf